CLINICAL TRIAL: NCT01818297
Title: SubQStim Pivotal Study: A Prospective, Randomized, Controlled Study to Evaluate the Safety and Efficacy of Subcutaneous Nerve Stimulation. Protocol 1666
Brief Title: Subcutaneous Nerve Stimulation for Failed Back Surgery Syndrome (FBSS) Patients
Acronym: SubQStim
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1666; G120146 (Other: FDA Protocol Number)
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Failed Back Surgery Syndrome; Post-laminectomy Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome; post laminectomy syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): Treatment settings of Medtronic PrimeAdvanced® neurostimulator system implant
  Interventions: Device: PrimeAdvanced® neurostimulator system
- Control (Other): Control settings of Medtronic PrimeAdvanced® neurostimulator system implant
  Interventions: Device: PrimeAdvanced® neurostimulator system

INTERVENTIONS:
Device: PrimeAdvanced® neurostimulator system — Neurostimulator and associated components

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Subcutaneous Nerve Stimulation (SQS) (also known as Peripheral Nerve Stimulation [PNS]) in the reduction of chronic, intractable post-surgical back pain in adults.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, randomized (1:1) parallel-group design.

ELIGIBILITY:
Key Inclusion Criteria:

* Have persistent back pain for at least 6 months
* Had back surgery at least 6 months ago
* Have tried pain medications and physical therapy
* Read and understand written English or Spanish
* Male or non-pregnant female. If female of child-bearing potential, and if sexually active, must be using a medically-acceptable method of birth control during study participation
* Willing and able to undergo surgical implant procedure, attend visits as scheduled, and comply with the study requirements
* Have an expected lifespan greater than 12 months

Key Exclusion Criteria:

* Have leg pain in addition to back pain.
* Currently enrolled in or plan to enroll in another drug and/or device study
* Have peripheral vascular disease, peripheral neuropathy, small-fiber neuropathy, or fibromyalgia
* Have an active systemic infection or are immunocompromised
* Will be exposed to diathermy or anticipate needing a full-body MRI scan
* Currently have an implantable cardiac pacemaker, defibrillator, or neurostimulator
* Treated with spinal cord stimulation, peripheral nerve stimulation, an intrathecal drug delivery system or requires additional back surgery

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Mandybur, MD, Principal Investigator — Mayfield Clinic, University of Cincinnati
Locations (27):
- United States (27):
  - Valley Pain Consultants, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Coastal Pain Research, Carlsbad, California
  - Pain Medicine Associates, Fountain Valley, California
  - Florida Pain Institute, Merritt Island, Florida
  - Advanced Medicine and Pain Management Research, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Willis Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - Comprehensive Pain and Rehabilitation, Pascagoula, Mississippi
  - Columbia Interventional Pain Center, LLP, Columbia, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - NYU Langone Medical Center, New York, New York
  - Mayfield Clinic, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Summa Western Reserve Hospital, Cuyahoga Falls, Ohio
  - DNA Advanced Pain Treatment Center, Greensburg, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Southern Spine Institute, Mt. Pleasant, South Carolina
  - Austin Pain Associates, Cedar Park, Texas
  - Space City Pain Specialists, Webster, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Wisconsin Health Center Surgery Center, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adult patients with chronic, intractable post-surgical back pain. First enrollment was in April 2013. Enrollment was suspended in September 2014 due to slow enrollment. The last subject visit was in March 2016. The planned enrollment was 323 subjects, with 218 randomized. Actual enrollment was 137 subjects with 62 randomized.
Pre-assignment Details: Of the 137 enrolled subjects, 62 were implanted and randomized. Of the 75 subjects who discontinued from the study prior to randomization, 54 did not meet inclusion/exclusion criteria, 12 withdrew consent or declined device implant, 3 discontinued due to study suspension, and 6 discontinued for other reasons.
Period: Blinded Phase (Randomization - 3 Months)
Arm/Group | Treatment | Control
Started | 32 | 30
Week 1 | 32 | 30
Week 6 | 32 | 29
Completed | 32 | 29
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Open Label Phase (3-12 Months)
Arm/Group | Treatment | Control
Started | 32 | 29
Completed | 14 | 19
Not Completed | 18 | 10
Not completed — Physician Decision | 1 | 0
Not completed — Early study closure | 17 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (13.1) | 59.8 (13.7) | 60.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 32 | 29 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 30 | 28 | 58
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62
Back pain [Mean (Standard Deviation); unit: units on a scale] — Average/typical back pain on a scale of 0 (no pain) - 10 (worst pain). Average of a back pain diary assessment.
  units on a scale | 6.77 (1.25) | 6.66 (0.88) | 6.71 (1.08)

OUTCOME MEASURES:

1. Primary Outcome: Number of Back Pain Responders (Subjects Who Achieve at Least a 50% Reduction in Average Back Pain With no Increase in Prescription Pain Medications) From Baseline to Month 3 Post-device Activation.
Description: Number of responders in Treatment and Control groups. Subjects reported typical back pain (0=no pain, 10=worst pain) during the Baseline (BL) and Blinded Phase (M3) periods. Percentage reduction in average back pain was calculated as (BL-M3)/BL. Subjects with at least a 50% reduction in average back pain between Baseline and Month 3, with no increase in prescribed pain medications, were considered responders.
Time Frame: Baseline to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 32 | 30
Participants | 9 | 5
Statistical Analysis 1: Comparison: Treatment vs Control; The original sample size estimate for the primary objective was based on the following assumptions: 109 subjects in each arm with a responder rate of 22% in the Control group and 40% in the Treatment group, and a one-sided α= 0.05 using a Z test with unpooled variance, would result in 90% power. Because the study terminated early, the actual sample size (32 in Treatment, 30 in Control) resulted in 47% power under the same assumptions; Test type: Superiority; p = 0.14, Z-test — Due to early termination, the study was insufficiently powered to test the primary objective. This analysis is exploratory and descriptive in nature and cannot be considered conclusive; The Z-test (using an unpooled standard deviation, without continuity correction) was used to test the difference in responder rates between groups; Risk Difference (RD) = 11.5, 95% CI 1-sided [lower limit -5.8], Standard Error of Mean 10.5 — The Estimation Parameter is the difference between the responder rates in the Treatment and Control groups. The difference is calculated as Treatment - Control. A positive number represents a higher responder rate in the Treatment group

2. Secondary Outcome: Functional Disability
Description: Compare the difference in average improvement in disability (as measured by Oswestry Disability Index (ODI)) from Baseline to Month 3 between the Treatment and Control groups. ODI ranges from 0% (no disability) -100% (greatest disability). Change is calculated as Baseline - Month 3 with a positive change indicating improvement in disability. Subjects with missing Baseline and/or Month 3 ODI assessments were counted as no change (Baseline - Month 3 = 0).
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 32 | 30
units on a scale | 9.8 (14.3) | 10.0 (12.1)

3. Secondary Outcome: Subject Satisfaction
Description: Compare difference in number of subjects satisfied with therapy between the Treatment and Control groups at Month 3. Subjects who reported they were very or somewhat satisfied with the therapy were counted as satisfied. Subjects with no satisfaction response were excluded from the analysis.
Time Frame: 3 months
Population: The analysis population includes all randomized subjects, with the exception of one subject in the Control group who did not have a satisfaction value. This subject was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 32 | 29
Participants | 25 | 22

4. Secondary Outcome: Quality of Life: Physical
Description: Compare the average change in quality of life (as measured by Short Form Health Survey (SF36 v2): Physical component score (PCS)) from Baseline to Month 3 between subjects in the Treatment and Control groups. The PCS ranges from 0 (worst possible physicial quality of life) to 100 (best possible physical quality of life). Change was calculated as Month 3 - Baseline, with a positive difference indicating improvement in physical quality of life. Subjects with missing Baseline and/or Month 3 SF-36: PCS assessments were counted as no change (Month 3 - Baseline = 0).
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 32 | 30
units on a scale | 3.6 (8.6) | 3.1 (7.1)

5. Secondary Outcome: Quality of Life: Mental
Description: Compare the average change in quality of life (as measured by Short Form Health Survey (SF36 v2): Mental component score (MCS)) from Baseline to Month 3 between subjects in the Treatment and Control groups. The MCS ranges from 0 (worst possible mental quality of life) to 100 (best possible mental quality of life). Change was calculated as Month 3 - Baseline, with a positive difference indicating improvement in mental quality of life. Subjects with missing Baseline and/or Month 3 SF-36: MCS assessments were counted as no change (Month 3 - Baseline = 0).
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 32 | 30
units on a scale | 1.9 (10.0) | 1.4 (9.6)

6. Secondary Outcome: Worst Back Pain
Description: Compare the average improvement in worst back pain from Baseline to Month 3 between the Treatment and Control groups. Subjects reported worst back pain (0 (no pain) - 10 (worst pain)) during the Baseline and Blinded Phase (Month 3) periods. Change was calculated as Baseline - Month 3, with a positive change indicating improvement in worst back pain.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 32 | 30
units on a scale | 2.7 (2.6) | 1.6 (1.9)

ADVERSE EVENTS:
Time Frame: The adverse events summarized by treatment arm are all adverse events that were collected during the Blinded Phase of the study (from Randomization through the Month 3 visit).
Description: There were 175.6 total months of subject follow-up during this time: 94.2 months in the Treatment group and 81.4 months in the Control group.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/32 | 0/30
Other Adverse Events (participants affected / at risk) | 11/32 | 8/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=32) | Control (N=30)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=32) | Control (N=30)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Implant site pain (General disorders) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Burning sensation (Nervous system disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to early study termination prior to completion of planned enrollment, the summaries describe the available data, and no conclusions can be made on the efficacy of the therapy based on the data available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restrictions on the PI allow for the sponsor to review results communications prior to public release and to embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to sponsor for review. The sponsor is also allowed to require changes for technical correctness and to protect confidential information, copyrightable or patentable material; and when reasonably requested, extend the embargo up to an additional 90 days.